CLINICAL TRIAL: NCT04138563
Title: Cardiac Output and Brain Perfusion and Architecture During Exercise in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Healthy, Age Matched Volunteers
Brief Title: Cerebral and Cardiac Blood Flow During Exercise in Patients With COPD
Acronym: REFLEX-COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 18063
Record Dates: First submitted 2019-10-17; First posted 2019-10-24 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: COPD; Cognitive Impairment
Keywords: Exercise; Magnetic Resonance Imaging; Cerebrovascular physiology; Cardiovascular physiology; Supine ergometric stepper
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood (plasma and serum) will be the only tissue collected. Upto 20 mls in total will be taken. some will be directly sent off for FBC, BNP and renal function. The rest of the serum will be aliquoted and stored for later research purposes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Participants with a pack year history of more than 10 pack years, diagnosed with COPD who have FEV1/FVC ratio of less than 0.7 AND FEV1 predicted value less than or equal to 60%.
- Control: Participants without a diagnosis of COPD who have a smoking history of more than 10 pack years

SUMMARY:
Heart disease and conditions related to the blood vessels are responsible for a large proportion (over a quarter) of the deaths in people with chronic obstructive pulmonary disease (COPD). The changes can also affect the smaller smaller blood vessels within the body, in particular the brain and the kidneys. This might be related to how the heart pumps and if it is under any pressure. Investigations performed at the University in healthy older volunteers demonstrated how the blood flows in the brain and heart during exercise. Exercise gently puts the whole body under some pressure and therefore exposes any weaker areas.

In this study the investigators are hoping to find out what happens to the blood flow in the brain and in the heart in patients who have COPD when they exercise and in the resting state. This will be compared to people of a similar age with a similar smoking history but without COPD. This will be examined using state of the art magnetic resonance imaging (MRI) and will allow us to assess whether changes in structure and function are related to this altered blood flow.

Our hypothesis is that COPD will cause a larger change in blood flow during exercise compared to the healthy volunteers and that reduced cardiorespiratory fitness will be associated with increased age related structural within the brain.

DETAILED DESCRIPTION:
The aim is to recruit 20 participants with COPD, who will be compared to 10 age and gender matched controls who also have a smoking history. The investigators aim for this number to complete the components of the study and therefore may have to over-recruit if some people drop out or are not eligible. The study elements are feasible, as the work extends a previous research study in healthy volunteers.

This research trial will consist of a medical screening visit and three investigation study visits spaced ideally one week apart. The investigation visits will begin within 6 (ideally within 4) weeks of the medical screening visit. The total duration of the study and screening visits should be 12 weeks maximum for each participant.

Screening visit:

If the participant expresses an interest in the clinical trial and wants to take part they will be invited (at a convenient time for them) to attend a medical screening visit located at the Nottingham City hospital. Here the investigator will discuss the research trial and answer any questions or concerns they might have regarding the research trial. The participant, if willing, will then be required to sign a consent form so that the screening procedures can begin, which include:

* Blood sample: Approximately a 20ml sample (4 teaspoons) taken from their arm, for further investigation including full blood count (FBC), brain natriuretic peptide (BNP) and kidney function.
* Questionnaires: 5 different questionnaires that ask about symptoms and how they affect daily life, a physical activity questionnaire, quality of life questionnaire and a MRI safety questionnaire.
* Spirometry: A simple blowing test to assess the participants' breathing which is performed three times.
* 12 lead ECG.
* a hand grip dynamometer to assess muscle strength
* timed up and go test: a test used to measure gait speed, where participants are asked to get up from a chair and walking to 3 meters and back, whilst being timed.
* to wear a step counter (Sensewear armband) for a week during waking hours to record steps.

Provided the ECG, step count (<10,000 steps) and other screening elements are ok, the participant will proceed to Study visit 1.

Strength and exercise test protocol:

The participant will be required to abstain from strenuous exercise for the 48 hours prior to the visit and also from alcohol and caffeine for 24 hours prior. Upon arrival they will perform a knee extension exercise so we can establish the muscle strength in the legs, specifically 3 maximal knee extensions with a 30 second rest in between. We will also measure fatigue by dong 20 extensions after a short break.

After a break they will then undergo an exercise test using an MRI compatible stepper device (Ergospect Cardiostepper) whilst in a supine position. This has been adapted to be similar to how they will exercise in the MRI scanner. Volunteers will start off stepping at a frequency of 65-70 steps a minute at the minimum workload and every 3 minutes get gradually a little harder until exhaustion is reached. Heart rate at rest and in response to exercise will be measured using a heart monitor. Participants will be given the option to have their expired gases also measured during exercise using a face mask, though this is not necessary if not tolerated. In the final minute of each workload we will take a finger prick test to measure the gases in the patients blood. A 3 lead ECG and oxygen saturation probe will be attached during exercise as safety measures and the protocol will be halted if oxygen saturation falls below 80% or if any relevant rhythm abnormalities are seen on the ECG trace.

The second study visit will be used to confirm the exercise and strength parameters measured in the first study visit.

MRI protocol:

A series of scans of the brain and heart will be taken at rest and then whilst stepping on the stepper machine within the MRI. The exercise will be at a steady state low level intensity determined by calculating the workload at which a fraction of maximum heart rate was achieved during first 2 study visits.

The MRI scan itself will take about ¾ hour but upto 2 hours is allowed for preparation and introducing the scan to the participant. The scanner is quite noisy and so the participant will wear ear defenders during the scan. Because the scanner is built around a large magnet, the participant will be instructed to remove all metal from their body, including jewellery. There is no radiation involved.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65-75 years old,
* >10 pack years smoking,
* FEV1/FVC <0.7 and FEV1<60% predicted (for COPD participants only)
* Sedentary lifestyle (<10,000 steps per day)
* Able to give informed consent
* Able to read, understand and communicate coherently in English

Exclusion Criteria:

* Doctor diagnosis of ischaemic heart disease or heart failure
* Doctor diagnosis of dementia or Alzheimers disease
* History of previous cerebrovascular disease (stroke or TIA) or malignancy
* Pregnancy or childbearing in the last 6 months
* Maintenance oral corticosteroids in the past 6 months
* Requirement for oral corticosteroids or antibiotics in the past 6 weeks
* Active arthritis or other muscular condition limiting exercise
* Surgical intervention in the last 12 weeks
* Long term oxygen therapy requirement
* Other formal current respiratory diagnosis
* Thyroid disease
* Diabetes Mellitus
* Neurological or cognitive impairment
* Significant physical disability
* Any other conditions in addition to the above that the investigators consider may affect study measurements or safety
* Inability to understand verbal and/or written explanation of the study requirements

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are recruiting participants within the Nottinghamshire region. Specifically for patients with COPD, we are targeting outpatient respiratory clinics at the Nottingham University Hospitals Trust, inpatient admissions due to COPD exacerbation at the Nottingham City Hospital, pulmonary rehabilitation groups and respiratory focus groups within Nottingham and patients on the Nottingham Respiratory Research Unit database.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Resting white and grey matter structural integrity | up to 12 weeks
  Grey and white matter volume (mm3) using the MRI MPRAGE sequences will be measured at rest
Cardiac structural integrity | up to 12 weeks
  Cardiac output (L/min) will be measured using the MRI sequence (Short axis Cine) at rest.
Cardiac structural integrity | up to 12 weeks
  Cardiac fibrosis (%) will be measured using the MRI MOLLI T1 sequence at rest.
Cardiac structural integrity | up to 12 weeks
  Myocardial strain (%) will be measured using the MRI cardiac tagging sequence at rest.
Whole body fat and muscle quantification | up to 12 weeks
  Whole body fat and muscle quantification (%) will be measured using the MRI whole body mdixon sequence at rest.
Aortic flow | up to 12 weeks
  Aortic flow (ml/min) will be measured during rest, low level steady-state exercise and following cessation of exercise and compared between COPD and age and gender matched controls
Cerebral blood flow | up to 12 weeks
  Cerebral blood flow (ml/min) will be measured during rest, low level steady-state exercise and following cessation of exercise and compared between COPD and age and gender matched controls
Cerebral perfusion | up to 12 weeks
  Cerebral artery perfusion (ml/100g/min) will be measured during rest, low level steady-state exercise and following cessation of exercise and compared between COPD and age and gender matched controls
Oxygen extraction fraction | up to 12 weeks
  Oxygen extraction fraction (%) will be derived from the difference between arterial and venous cerebral oxygenation measured via TRUST MRI scan sequence during rest, low level steady-state exercise and following cessation of exercise and compared between COPD and age and gender matched controls

SECONDARY OUTCOMES:
Muscle isometric strength (MVC) | up to 6 weeks
  Isometric muscle torque of the quadriceps (Nm) assessed using the cybex dynamometer
Muscle isokinetic fatigue | up to 6 weeks
  Fatiguability test of the quadriceps (Nm) assessed using the cybex dynamometer
Quality of life (SGRQ) | 1 week
  Assessed using the St Georges Respiratory Questionnaire. min value: 0, max value: 84, higher score means worse outcome
Physical activity level (IPAQ Physical activity questionnaire) | 1 week
  Assessed using the International Physical activity questionnaire. min value: 0, max value: 66000, higher score means better outcome
Montreal Cognitive Assessment (MoCA) cognition level | 1 week
  Assessed using the Montreal cognitive assessment questionnaire. min value: 0, max value: 30, higher score means better outcome
Hospital anxiety and depression scale (HADS) | 1 week
  min value: 0, max value: 21, higher score means worse outcome
Hand grip strength | 1 week
  Composite of hand grip strength (Kg), measured by a hand held dynamometer,
Timed up and go test | 1 week
  Timed up and go test (seconds) will be measured to assess degree of frailty.
Serum markers of inflammation for research purposes (likely to include IL-1, IL-6, and TNFα) | 1 week
  Blood test
Heart rate response to exercise | up to 6 weeks
  Heart rate response (Beats per minute) will be measured at rest and during incremental exercise to assess cardio-respiratory fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Bolton, Principal Investigator — NIHR Nottingham Biomedical Research Centre Respiratory theme, University of Nottingham
Locations (1):
- NIHR Nottingham BRC Respiratory Theme, University of Nottingham and NUH Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McGarvey LP, John M, Anderson JA, Zvarich M, Wise RA; TORCH Clinical Endpoint Committee. Ascertainment of cause-specific mortality in COPD: operations of the TORCH Clinical Endpoint Committee. Thorax. 2007 May;62(5):411-5. doi: 10.1136/thx.2006.072348. Epub 2007 Feb 20. PMID 17311843
- [Background] Sabit R, Bolton CE, Edwards PH, Pettit RJ, Evans WD, McEniery CM, Wilkinson IB, Cockcroft JR, Shale DJ. Arterial stiffness and osteoporosis in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2007 Jun 15;175(12):1259-65. doi: 10.1164/rccm.200701-067OC. Epub 2007 Mar 15. PMID 17363772
- [Background] John M, Hussain S, Prayle A, Simms R, Cockcroft JR, Bolton CE. Target renal damage: the microvascular associations of increased aortic stiffness in patients with COPD. Respir Res. 2013 Mar 5;14(1):31. doi: 10.1186/1465-9921-14-31. PMID 23497267
- [Background] Blair SN, Kohl HW 3rd, Paffenbarger RS Jr, Clark DG, Cooper KH, Gibbons LW. Physical fitness and all-cause mortality. A prospective study of healthy men and women. JAMA. 1989 Nov 3;262(17):2395-401. doi: 10.1001/jama.262.17.2395. PMID 2795824
- [Background] Erickson KI, Leckie RL, Weinstein AM. Physical activity, fitness, and gray matter volume. Neurobiol Aging. 2014 Sep;35 Suppl 2:S20-8. doi: 10.1016/j.neurobiolaging.2014.03.034. Epub 2014 May 14. PMID 24952993